CLINICAL TRIAL: NCT07367100
Title: A Prospective, First in Human Pivotal Study to Evaluate the Adaptive Tip Catheter Used to Treat Acute Ischemic Stroke Patients During Mechanical Thrombectomy
Brief Title: A Pivotal Study Evaluating Safety and Effectiveness of Adaptative Tip Catheter in Patients With Acute Ischemic Stroke
Acronym: PHAST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neuravi Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNV202304
Record Dates: First submitted 2026-01-16; First posted 2026-01-26 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Ischemic Stroke
Keywords: Large Vessel Occlusion; Acute Ischemic Stroke; Mechanical Thrombectomy
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adaptive Tip Catheter (ATC) (Experimental): The ATC will be used alone (direct aspiration) as the first attempted device/technique for mechanical thrombectomy in the anterior circulation in patients during the first three passes or until final reperfusion, if less than three passes are needed. Patients will be followed over 90 days post procedure.
  Interventions: Procedure: Adaptive Tip Catheter

INTERVENTIONS:
Procedure: Adaptive Tip Catheter — Patients will undergo mechanical thrombectomy using ATC.

SUMMARY:
The purpose of this study is to assess the safety and the effectiveness of the Adaptive Tip Catheter (ATC) used as a first line direct aspiration thrombectomy technique for patients suffering of an acute ischemic stroke.

ELIGIBILITY:
Inclusion criteria:

* Age greater than or equal to (>=) 18 years, less than or equal to (<=) 90 years, at the time of consent
* Signs and symptoms consistent with the diagnosis of acute ischemic stroke in the anterior circulation that can be treated with endovascular thrombectomy approaches
* Endovascular treatment can be initiated (defined as access puncture) within 24 hours from time last known well
* Baseline National Institutes of Health Stroke Scale (NIHSS) score >= 6
* A signed and dated Informed Consent Form (ICF) or Investigator Statement for emergency procedure (as allowed according to country regulations and approved by EC) has been obtained

Exclusion criteria:

* Known pregnancy, as evidenced by positive pregnancy test for women of childbearing potential or breast feeding
* Life expectancy less than (<) 90 days prior to stroke onset
* Known hemorrhagic diathesis disorder, coagulation factor deficiency or oral anticoagulant therapy with known International Normalized Ratio (INR) greater than (>) 3.0
* Clinical symptoms and/or CT/MRI evidence suggestive of bilateral stroke or stroke in multiple vascular territories, defined as occlusions in more than one vessel not downstream from each other (for example, bilateral anterior circulation, anterior/posterior circulation)
* Clinical history, past imaging or clinical judgement suggest that the intracranial occlusion is chronic
* Computed Tomography/ Magnetic Resonance Imaging (CT/MRI) evidence of recent/fresh hemorrhage
* Baseline CT or MRI showing mass effect
* Currently participating in an investigational (drug, device, etc.) clinical trial that may confound study endpoints. Patients in observational, natural history, and/or epidemiological studies not involving intervention are eligible
* Cerebral catheter angiographic evidence of pre-existing arterial disease, that potentially impacts treatment and/or outcome (for example, vasculitis)
* Any occlusion or stenosis that limits device access to the target area (for example, carotid dissection, tandem occlusions) or requiring acute stenting to achieve access
* Cerebral catheter angiographic evidence of multiple cerebrovascular occlusions, defined as occlusions in more than one vessel not downstream from each other (for example, bilateral anterior circulation, anterior/posterior circulation)
* Excessive vascular access tortuosity that will likely prevent endovascular access with the adaptive tip catheter (ATC)
* Baseline expanded thrombolysis in cerebral infarction (eTICI) > 1

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2026-02-02 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Third Pass Reperfusion Assessed by Independent Imaging Core Lab | Intraoperative
  Successful achievement of the third pass reperfusion is defined as achieving an Expanded Thrombolysis in Cerebral Infarction (eTICI) score of 2b50 or greater using no more than three passes with the study device in the target vessel, and without any rescue therapy.

SECONDARY OUTCOMES:
First Pass Reperfusion | Intraoperative
  Successful achievement of the first pass reperfusion is defined as achieving an eTICI score of 2c or greater, as determined by the independent imaging core lab, with one pass of the study device in the target vessel, and without any rescue therapy.
Final Procedural Reperfusion | Intraoperative
  Successful achievement of the final procedural reperfusion is defined as achieving a final (end of procedure) eTICI score of 2b50 or greater in the target vessel as determined by the independent imaging core lab.
Modified Rankin Scale (mRS) Score of 0-2 at 90 days Post-Procedure | At 90 days post-procedure
  Percentage of patients with mRS score of 0-2 at 90 days or no change from baseline if pre-ictal mRS greater than (>) 2 will be reported.
Vessel Damage | At 90 days post-procedure
  Number of patients with perforation or dissection in the blood vessel known to be related to or possibly related to the study device will be reported.
All-Cause Mortality | At 90 days post-procedure
  All mortality regardless of causes at 90 days post-procedure will be reported.
Symptomatic Intracranial Hemorrhage (sICH) at 24 hours | At 24 hours after intervention
  sICH is defined as a new intracranial hemorrhage as detected by brain imaging, measured 24 hours after intervention associated with any of the following: greater than or equal to (>=) 4 points total National Institutes of Health Stroke Scale (NIHSS) at the time of diagnosis compared to immediately before worsening; >= 2 point in one NIHSS category; leading to intubation/hemicraniectomy/external ventricular drain (EVD) placement or other major medical/surgical intervention or absence of alternative explanation for deterioration.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Cognard, MD-PhD, Principal Investigator — CHU Toulouse - Hôpital, Purpan, Toulouse France
Locations (15):
- Belgium (3):
  - UZ Antwerpen, Edegem
  - Ghent University Hospital, Ghent
  - Universitair Ziekenhuis Leuven, Leuven
- France (5):
  - CHU Bordeaux, Bordeaux
  - CHU Nantes, Nantes
  - CHU Pitie Salpetriere, Paris
  - Centre Hospitalier Universitaire de Toulouse - Hopital Purpan, Toulouse
  - CHRU de Tours, Tours
- Germany (4):
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitatsklinikum Schleswig Holstein Kiel, Kiel
  - Universitaetsmedizin Mainz, Mainz
  - Stadtisches Klinikum Solingen gemeinnutzige GmbH, Solingen
- Beaumont Hospital, Dublin, Ireland
- Netherlands (2):
  - VUMC Amsterdam, Amsterdam
  - Maastricht University Medical Centre, Maastricht

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu.
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency